CLINICAL TRIAL: NCT06830772
Title: Acute Physiological and Psychological Responses to Virtual and Mixed Reality Exergaming During Workplace Breaks: An Exploratory Crossover Trial
Brief Title: Affective and Physiological Outcomes of Virtual and Mixed Reality Workplace Exergames
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Abdullah Kayhan, Research Assistant, Akdeniz University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 21012025-02-47
Record Dates: First submitted 2025-02-12; First posted 2025-02-17 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Exergame; Active Video Games (AVG); Virtual Reality; Mood Changes
Keywords: exergame; active video game; virtual exergame
MeSH Terms: interventions — Exergaming

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Virtual Reality Exergame (VR-EX) (Experimental): Participants will engage in a Virtual Reality (VR)-based exergame session using the PowerBeatsVR application. The session will include rhythm-based exercises, such as punching targets and dodging obstacles, aimed at promoting physical activity during a short break in the workplace.
  Interventions: Other: Experimental
- Mixed Reality Exergame (MR-EX) (Active Comparator): Participants will engage in a Mixed Reality (MR)-based exergame session using the PowerBeatsVR application in MR mode. This condition allows participants to interact with virtual elements while maintaining awareness of their physical surroundings.
  Interventions: Other: Active comparator
- Passive Rest (PR) (No Intervention): Participants will remain seated in a quiet room for the same duration as the VR and MR sessions. During this time, they will be asked to rest without engaging in any physical activity. Talking, using mobile devices, or interacting with others will not be allowed to ensure a consistent resting condition across participants.

INTERVENTIONS:
Other: Experimental — Virtual Reality Exergame (VR) Participants will engage in a 5-minute fully immersive Virtual Reality (VR) exergame session using the PowerBeatsVR application. This intervention takes place in a virtual environment where participants perform rhythm-based physical activities such as punching targets and dodging obstacles. The VR session isolates participants from their real-world surroundings, offering a highly immersive experience designed to promote physical activity and assess its physiological and psychological effects.
  Other Names: Virtual Reality Exergame
  Arms: Virtual Reality Exergame (VR-EX)
Other: Active comparator — Mixed Reality Exergame (MR) Participants will engage in a 5-minute Mixed Reality (MR) exergame session using PowerBeatsVR in MR mode. Unlike VR, this intervention integrates virtual elements into the real-world environment, allowing participants to maintain awareness of their physical surroundings while interacting with digital content. This hybrid experience reduces the risk of cybersickness while providing a practical approach for workplace settings.
  Other Names: Mixed Reality Exergame
  Arms: Mixed Reality Exergame (MR-EX)

SUMMARY:
The aim of this study was to compare the acute effects of virtual reality (VR) and mixed reality (MR) based exergame practices on physical and psychological health indicators during micro-breaks among university administrative staff. The main research questions aimed to be answered are:

1. How does VR exergame and MR exergame affect physical health indicators such as heart rate and perceived exertion in university administrative staff?
2. How does MR exergame with VR exergame affect the mood of university administrative staff?
3. How does MR exergame with VR exergame affect the enjoyment of exercise and gaming experience of university administrative staff?

Researchers will compare passive rest with VR Exergame and MR exergame to see if VR and MR sessions improve physical and psychological outcomes compared to passive rest.

Participants will: Sit quietly in a designated room for 5 minutes without engaging in any physical activity. Avoid talking, using mobile devices, or interacting with others during the rest session to ensure consistent conditions for all participants.

DETAILED DESCRIPTION:
Using a randomized crossover design, participants will experience three different conditions: VR-based exergames, MR-based exergames, and passive rest. Each condition will be performed on separate days, with a minimum of 48 hours between sessions to prevent carryover effects.

The primary outcomes will include mood states, heart rate, and perceived exertion. These measures will help assess the immediate physical and psychological responses to the interventions.

The secondary outcomes will focus on exercise enjoyment and overall gaming experience, evaluating the subjective experience and engagement levels during VR and MR exergaming sessions.

The intervention will be delivered through PowerBeatsVR, a rhythm-based exergame that requires physical movements such as dodging obstacles and throwing punches. VR and MR modes will be compared to determine their effectiveness in promoting physical activity and improving mood during short breaks in a workplace setting. The passive rest condition will serve as a baseline for comparison.

This study addresses the growing interest in workplace wellness strategies by exploring the potential of VR and MR exergames in reducing sedentary behavior and enhancing mental well-being in work environments.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over
* Being suitable for physical activity according to PAR-Q test
* Not exercising for 30 minutes 3 days a week
* Not having used VR/MR technologies before

Exclusion Criteria:

* People with epilepsy, vertigo or neurological diseases
* Use of antidepressants or similar medication
* Individuals with high Physical Activity Level (IPAQ)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2025-02-26 (Actual); Primary Completion 2025-04-11 (Actual); Study Completion 2025-04-11 (Actual)

PRIMARY OUTCOMES:
Mood State | Baseline and immediately post-intervention (within 5 minutes after the session)
  Participants' mood states will be assessed before and after each session using the Brunel Mood Scale (BRUMS). The scale consists of 24 items and 6 subscales rated on a 5-point Likert scale (0 = Not at all, 4 = Extremely).
Heart Rate | Baseline, during intervention, and immediately post-intervention (within 5 minutes after the session)
  Heart rate will be measured using a POLAR H20 heart rate monitor at baseline, during the session, and immediately post-intervention. Data will be recorded in real time through the Polar Flow application to assess physical activity intensity.
Perceived Exertion | Baseline and immediately post-intervention (within 5 minutes after the session)
  Perceived exertion will be evaluated using the Borg Rating of Perceived Exertion (RPE) Scale (6-20) after each session. This scale measures subjective physical effort perception and is widely used for assessing exercise intensity.

SECONDARY OUTCOMES:
Exercise Enjoyment | Immediately post-intervention (within 5 minutes after the session)
  Exercise enjoyment will be assessed using the Physical Activity Enjoyment Scale (PACES). The short form of the scale consists of 5 items rated on a 7-point bipolar Likert scale. Higher scores indicate greater enjoyment of the physical activity experience.
Game Experience (Dominance and Absorption) | Immediately post-intervention (within 5 minutes after the session)
  The gaming experience will be evaluated using the Gameful Experience Scale (GAMEX), focusing on the subscales of Dominance and Absorption. These subscales measure the participant's sense of control and engagement during the gaming session, with responses rated on a 5-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Tennur Yerlisu Lapa, Study Director — Akdeniz University
Locations (1):
- Akdeniz University, Konyaalti, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No